CLINICAL TRIAL: NCT06686797
Title: A PHASE 1, RANDOMIZED STUDY WITH DOUBLE-BLIND AND SPONSOR-OPEN, PLACEBO-CONTROLLED SINGLE- AND MULTIPLE-DOSE ESCALATION TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF PF-08049820 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-08049820 Are Tolerated and Act in the Body in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C6231001; NCT06686797 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind, sponsor-open study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A: Cohort 1 (Experimental): Up to 4 dosing periods in healthy adult participants. Each period consists of a single dose of PF-08049820 or placebo.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part A: Cohort 2 (Experimental): Up to 4 dosing periods in healthy adult participants. Each period consists of a single dose of PF-08049820 or placebo.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part A: Cohort 3 (Experimental): One dosing period with a single dose of PF-08049820 or placebo in healthy adult Japanese participants.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part B: Cohort 4 (Experimental): One dosing period with multiple doses of PF-08049820 or placebo in healthy adult participants.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part B: Cohort 5 (Experimental): One dosing period with multiple doses of PF-08049820 or placebo in healthy adult participants.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part B: Cohort 6 (Experimental): One dosing period with multiple doses of PF-08049820 or placebo in healthy adult participants.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part B: Cohort 7 (Experimental): One dosing period with multiple doses of PF-08049820 or placebo in healthy adult participants.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part C: Cohort 8 (Experimental): One dosing period with a single dose of PF-08049820 or placebo in healthy adult participants.
  Interventions: Drug: PF-08049820; Drug: Placebo
- Part C: Cohort 9 (Experimental): One dosing period with a single dose of PF-08049820 or placebo in healthy adult participants.
  Interventions: Drug: PF-08049820; Drug: Placebo

INTERVENTIONS:
Drug: PF-08049820 — Oral solution/suspension for Part A (Cohorts 1 to 3). Tablets for Parts B and C (Cohorts 4 to 9).
Drug: Placebo — Oral solution/suspension for Part A (Cohorts 1 to 3). Tablets for Parts B and C (Cohorts 4 to 9).

SUMMARY:
The purpose of this study is to learn about the safety of the study medicine called PF-08049820 in healthy adults. The study will also see:

* how the body processes the study medicine and
* if food affects the amount of study medicine in the blood.

The study medicine is developed for the treatment of moderate to severe atopic dermatitis, also known as eczema. People with this condition may have severe itching and rashes on the skin.

The study is seeking participants who:

1. Are males or females who can no longer have children,
2. Are 18 to 65 years old,
3. Have a body mass index (BMI) of 16 to 32 kilograms per meter squared and a total body weight of more than 50 kilograms (110 pounds).

   For group or cohort 3 only:
4. Have 4 biological Japanese grandparents who were born in Japan.

The study has three parts: Part A, Part B and Part C.

Part A consists of 3 groups (also known as "cohorts"). In Cohorts 1 and 2, there may be up to four dosing periods. During each dosing period, participants will take a single dose of the study medicine or placebo as liquid by mouth with or without food at the study clinic. A placebo does not have any medicine in it but looks just like the medicine being studied. The participants will stay at the study clinic for about 8 days and then can go home. During this time, the study team will observe the participants and take some urine and blood samples to test the level of the study medicine. The participants will return to the study clinic up to three more times to complete up to four dosing periods separated by at least 2 weeks. The participants will take increasing amounts of study medicine during each dosing period. After completion of the final dosing period, the participants will receive a follow-up telephone call about a month later. Cohort 3 consists of one dosing period and will enroll participants who have 4 biological Japanese grandparents who were born in Japan. Participants will be checked as described above and will receive a follow-up telephone call about one month after the last dose of study medicine or placebo.

Part B has 4 cohorts (Cohorts 4 to 7), each consisting of one dosing period. In all cohorts, participants will take multiple doses of the study medicine or placebo as tablets by mouth at the study clinic. Part C has two cohorts (Cohort 8 and 9), each consisting of one dosing period. In both cohorts, participants will take a single dose of the study medicine or placebo as tablets by mouth at the study clinic. Participants will be checked as described above and will receive a follow-up telephone call about one month after the last dose of study medicine or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females who can no longer have children.
2. Body mass index (BMI) of 16-32 kg/m2; and a total body weight >50kg (110 lb.). Japanese participants only: a total body weight >45 kg is acceptable.

   Cohort 3 only:
3. Have 4 biological Japanese grandparents who were born in Japan

Exclusion criteria

1. Evidence or history of clinically significant medical conditions.
2. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb).
3. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
4. Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline up to Day 35 of last dosing period for Parts A and C and up to Day 45 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Number of Participants With Serious Adverse Events (SAEs) | Baseline up to Day 35 of last dosing period for Parts A and C and up to Day 45 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to Day 21 of last dosing period for Parts A and C and up to Day 31 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Day 21 of last dosing period for Parts A and C and up to Day 31 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings | Baseline up to Day 21 of last dosing period for Parts A and C and up to Day 31 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | Baseline up to Day 8 of last dosing period for Parts A and C
  Part A (Cohorts 1 to 3) Part C (Cohorts 8 and 9)
Area under the curve from time zero to end of dosing interval (AUCtau) | Baseline up to Day 13 for Part B
  Part B (Cohorts 4 to 7)
Maximum observed plasma concentration (Cmax) | Baseline up to Day 8 of last dosing period for Parts A and C and up to Day 13 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Time to reach maximum observed plasma concentration (Tmax) | Baseline up to Day 8 of last dosing period for Parts A and C and up to Day 13 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Area under the curve from time zero to extrapolated infinite time (AUCinf) if data permit | Baseline up to Day 8 of last dosing period for Parts A and C and up to Day 13 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Plasma decay half-life (t1/2) if data permit | Baseline up to Day 8 of last dosing period for Parts A and C and up to Day 13 for Part B
  Part A (Cohorts 1 to 3) Part B (Cohorts 4 to 7) Part C (Cohorts 8 and 9)
Amount of unchanged drug recovered in urine during dosing interval (Aetau) | Baseline up to Day 10 for Part B
  Part B (Cohorts 4 to 7)
Percent of dose recovered in urine as unchanged drug over dosing interval (Aetau%) | Baseline up to Day 10 for Part B
  Part B (Cohorts 4 to 7)
Renal clearance (CLr) | Baseline up to Day 10 for Part B
  Part B (Cohorts 4 to 7)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6231001